CLINICAL TRIAL: NCT04704349
Title: Latest Imaging SPECT System Evaluation Phase 1
Acronym: LISSE1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHRO-2019-12
Record Dates: First submitted 2021-01-06; First posted 2021-01-11 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Rheumatic Disease; Neoplasms; Parathyroid Diseases; Pulmonary Embolism; Heart Diseases; Thyroid Diseases; Kidney Diseases; Dementia; Parkinsonian Disorders
Keywords: Gamma camera; whole body scan; scintigraphy
MeSH Terms: conditions — Rheumatic Diseases; Neoplasms; Parathyroid Diseases; Pulmonary Embolism; Heart Diseases; Thyroid Diseases; Kidney Diseases; Dementia; Parkinsonian Disorders

STUDY DESIGN:
Intervention Model Description: All patients will undergo scintigraphy on 2 distinct devices and the images obtained will be compared.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Scintigraphy acquisitions (Experimental): All patients will undergo scintigraphy on 2 distinct devices and the images obtained will be compared.
  Interventions: Radiation: Scintigraphy

INTERVENTIONS:
Radiation: Scintigraphy — The scintigraphy of the patients will be carried out on 2 distinct devices and the images obtained will be compared.

SUMMARY:
Monocentric study for the evaluation of a whole body CZT scintigraphy system.

DETAILED DESCRIPTION:
Monocentric evaluation of performances and clinical interest of a whole body scintigraphic acquisition system with CZT digital detectors. Comparison of image quality and resolution of the new system compared to a reference one, on phantoms and during the acquisition of a wide variety of examinations.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to our Nuclear Medicine department for bone, cardiac, pulmonary, thyroid, parathyroid, renal or cerebral perfusion scintigraphy or to DaTSCAN.

Exclusion Criteria:

* Under 18 years old patients.
* Pregnant women or at risk of pregnancy.
* Patients under guardianship
* Painful patient (EVA>4)
* Patients in whom a standard examination is not feasible (agitation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Rate of images with a score greater than or equal to 4 | Day 0
  Rate of images obtaining a score greater than or equal to 4 in visual image quality analysis on a 5-point LIKERT scale.

SECONDARY OUTCOMES:
collimator performance | Day 0
  Physical measurements of collimator performance on test object.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles METRARD, Dr, Principal Investigator — CHR Orléans
Locations (1):
- CHR d'Orleans, Orléans, France

REFERENCES:
- [Background] Garcia EV, Faber TL, Esteves FP. Cardiac dedicated ultrafast SPECT cameras: new designs and clinical implications. J Nucl Med. 2011 Feb;52(2):210-7. doi: 10.2967/jnumed.110.081323. Epub 2011 Jan 13. PMID 21233190
- [Background] Garcia EV. Are SPECT measurements of myocardial blood flow and flow reserve ready for clinical use? Eur J Nucl Med Mol Imaging. 2014 Dec;41(12):2291-3. doi: 10.1007/s00259-014-2924-2. No abstract available. PMID 25311927
- [Background] Slomka PJ, Berman DS, Germano G. New cardiac cameras: single-photon emission CT and PET. Semin Nucl Med. 2014 Jul;44(4):232-51. doi: 10.1053/j.semnuclmed.2014.04.003. PMID 24948149
- [Background] Bani Sadr A, Testart N, Tylski P, Scheiber C. Reduced Scan Time in 123I-FP-CIT SPECT Imaging Using a Large-Field Cadmium-Zinc-Telluride Camera. Clin Nucl Med. 2019 Jul;44(7):568-569. doi: 10.1097/RLU.0000000000002554. PMID 30932983
- [Background] Salerno M, Beller GA. Noninvasive assessment of myocardial perfusion. Circ Cardiovasc Imaging. 2009 Sep;2(5):412-24. doi: 10.1161/CIRCIMAGING.109.854893. No abstract available. PMID 19808630
- [Background] Mowatt G, Vale L, MacLeod A. Systematic review of the effectiveness of home versus hospital or satellite unit hemodialysis for people with end-stage renal failure. Int J Technol Assess Health Care. 2004 Summer;20(3):258-68. doi: 10.1017/s0266462304001060. PMID 15446754
- [Background] Loong CY, Anagnostopoulos C. Diagnosis of coronary artery disease by radionuclide myocardial perfusion imaging. Heart. 2004 Aug;90 Suppl 5(Suppl 5):v2-9. doi: 10.1136/hrt.2003.013581. No abstract available. PMID 15254003
- [Background] Roach PJ, Gradinscak DJ, Schembri GP, Bailey EA, Willowson KP, Bailey DL. SPECT/CT in V/Q scanning. Semin Nucl Med. 2010 Nov;40(6):455-66. doi: 10.1053/j.semnuclmed.2010.07.005. PMID 20920635
- [Background] Valotassiou V, Malamitsi J, Papatriantafyllou J, Dardiotis E, Tsougos I, Psimadas D, Alexiou S, Hadjigeorgiou G, Georgoulias P. SPECT and PET imaging in Alzheimer's disease. Ann Nucl Med. 2018 Nov;32(9):583-593. doi: 10.1007/s12149-018-1292-6. Epub 2018 Aug 20. PMID 30128693